CLINICAL TRIAL: NCT07054632
Title: Efficacy and Safety of Gene Therapy rAAV-RPE65 (LX101) in Biallelic RPE65 Mutation-associated Inherited Retinal Dystrophy: a Phase III, Multicenter, Randomized Controlled Trial (STAR)
Brief Title: Efficacy and Safety of LX101 for Inherited Retinal Dystrophy Associated With RPE65 Mutations
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Innostellar Biotherapeutics Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: INNOSTELLAR-LX101-1 (phase 2)
Record Dates: First submitted 2025-06-27; First posted 2025-07-08 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-07

CONDITIONS: Inherited Retinal Dystrophy Associated With RPE65 Mutations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental)
  Interventions: Genetic: LX101
- Control group (No Intervention)

INTERVENTIONS:
Genetic: LX101 — Subretinal administration of LX101 to the study eye
  Arms: Intervention group

SUMMARY:
The purpose of the study is to evaluate the efficacy and safety of LX101 in subjects with biallelic RPE65 mutation-associated inherited retinal dystrophy. This is an open-label, multicenter, randomized controlled Phase III clinical trial. Subjects were randomly assigned in a 1:1 ratio to either the intervention group or the control group. Subjects in the intervention group received subretinal injection of LX101, while those in the control group received no treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject and/or their guardian signing a written informed consent.

Diagnosed with biallelic RPE65 mutation-associated inherited retinal dystrophy.

Subjects are 6 years of age or older.

Visual acuity of ≤ 20/63 or visual field less than 20 degrees in the eye to be injected.

Exclusion Criteria:

* Prior gene therapy for IRD and other hereditary eye diseases.

Pre-existing eye conditions that would interfere with interpretation of study endpoints.

Active intraocular or periocular infections in the study eye.

Lacking of sufficient surviving retinal cells.

Prior ocular surgery within six months.

Complicating systemic diseases or clinically significant abnormal baseline laboratory values.

Pre-existing systemic diseases that should not discontinue the use of any retinal toxic compounds.

Complicating systemic diseases or clinically significant abnormal baseline laboratory values.

Min Age: 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-09-13 (Actual); Primary Completion 2025-08-13 (Estimated); Study Completion 2029-08 (Estimated)

PRIMARY OUTCOMES:
Mobility Test | 12 months
  Changes in functional vision from baseline, determined by mobility test score

SECONDARY OUTCOMES:
Full-field Light Sensitivity Threshold (FST) Test | 6 months、12 months
  Changes in light sensitivity from baseline, assessed by FST in log cd.s/m2
Visual Acuity | 6 months、12 months
  Changes in visual acuity from baseline, based on the ability to read letters using the Early Treatment Diabetic Retionpathy Study (ETDRS) chart
Mobility Test | 6 months
  Changes in functional vision from baseline, determined by mobility test score
Safety: Incidence of adverse events (AEs) and serious adverse events (SAEs) | 12 months
  Incidence of ocular and non-ocular AEs and SAEs following LX102 subretinal injection

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Zhongshan Ophthalmic Center, Sun Yat sen University, Guangzhou, Guangdong
  - Southwest Hospital of AMU, Chongqing
  - Shanghai General Hospital, Shanghai
  - Tianjin Medical University Ophthalmology Hospital, Tianjin